CLINICAL TRIAL: NCT07213453
Title: Evaluation of the Accuracy of Temporary Laminate Restorations Designed Using Two Different Digital Smile Design Workflows: A Pilot Study
Brief Title: Accuracy of Temporary Laminate Restorations With Digital Workflows
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Marmara Prostho Murat Feriz
Record Dates: First submitted 2025-09-22; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Esthetics, Dental
Keywords: Digital dentistry; Laminate veneer restorations; Esthetics; Accuracy; Digital Smile Design

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smilecloud Workflow (Experimental): Six laminate veneer restorations (canine-to-canine) designed via SmileCloud, beginning with 2D photographs and converted into 3D models before fabrication.
  Interventions: Device: Digital Smile Design
- Smile Creator Workflow (Experimental): Six laminate veneer restorations (canine-to-canine) designed directly in 3D using Smile Creator with integration of intraoral scans and extraoral photographs.
  Interventions: Device: Digital Smile Design

INTERVENTIONS:
Device: Digital Smile Design — Digital Smile Design workflows used for virtual planning and fabrication of laminate veneer restorations.

SUMMARY:
This pilot clinical study investigates the dimensional accuracy of temporary laminate veneer restorations designed using two distinct digital smile design (DSD) workflows. Five healthy volunteers with intact maxillary anterior dentition and good oral hygiene were enrolled at Marmara University, Faculty of Dentistry. Two digital workflows were compared: (1) a 2D-to-3D transformation approach using SmileCloud, where extraoral photographs are initially used for two-dimensional planning before conversion to 3D models, and (2) a direct three-dimensional design workflow using Exocad Smile Creator, which integrates intraoral scans and extraoral photographs at the initial stage. A total of 60 provisional laminate veneers were virtually designed and fabricated using stereolithography (SLA) 3D printing technology with ceramic-based resin. Dimensional measurements of mesiodistal tooth widths, inciso-gingival lengths, and intercanine distances were obtained from both digital designs and printed restorations. Statistical analysis compared the accuracy of virtual-to-physical transfer in both workflows. The findings aim to provide preliminary evidence on the reliability of digital smile design approaches for esthetic treatment planning and fabrication of temporary restorations.

DETAILED DESCRIPTION:
Aesthetic dentistry increasingly emphasizes minimally invasive procedures that integrate objective clinical standards with patients' esthetic expectations. Porcelain laminate veneers are one of the most widely accepted restorative approaches for enhancing smiles while preserving tooth structure. Provisional restorations play a central role in this process by offering a tangible preview of the anticipated outcome before irreversible treatment is performed. With the advancement of digital technologies, diagnostic mock-ups can now be generated virtually, converted into STL files, and fabricated with high precision using 3D printing. Within this context, digital smile design (DSD) has become a systematic tool that enhances communication, improves diagnostic accuracy, and supports predictable esthetic outcomes.

The present pilot study evaluates two distinct DSD workflows with the goal of assessing their dimensional accuracy in translating virtual designs into physical provisional restorations. Smilecloud initiates the planning process with two-dimensional photographic data. It automatically generates a smile frame based on facial references and provides a curated library of esthetic tooth shapes that can be customized. Once finalized, the 2D design is converted into a 3D model, which is later superimposed onto intraoral scans using dental CAD software. This workflow offers advantages for rapid case visualization and patient communication; however, its reliance on 2D projections may introduce errors in representing transverse dental relationships.

In contrast, Exocad Smile Creator employs a direct 3D workflow, integrating intraoral scans and extraoral photographs from the beginning. This enables precise alignment of dental arches with facial reference lines, allowing clinicians to make real-time adjustments. By eliminating intermediate data conversions, this approach is expected to minimize error propagation and provide greater dimensional fidelity.

Five volunteers aged 18-45 years with intact anterior dentition and good periodontal health were recruited. Standardized photographic records were obtained, and intraoral digital impressions were recorded with the 3Shape TRIOS 3 scanner. For each participant, six laminate veneer restorations were digitally designed in both workflows, resulting in a total of 60 provisional veneers.

All virtual designs were exported as STL files and fabricated with a stereolithography (SLA) 3D printer using a ceramic-based resin. Post-processing included rinsing in isopropyl alcohol, UV curing, and polishing. Dimensional measurements were performed both digitally and on fabricated restorations using a high-precision digital caliper. Parameters included mesiodistal tooth widths, inciso-gingival lengths, and intercanine arch width.

Statistical analysis assessed differences between virtual designs and physical restorations. Results indicated that vertical parameters showed no significant discrepancies across workflows. However, intercanine width was significantly underestimated in the 2D-based Smilecloud designs. Direct 3D workflows demonstrated close agreement between digital and physical outcomes.

This study demonstrates that both Smilecloud and Smile Creator can produce clinically acceptable provisional restorations, but dimensional fidelity is enhanced when a direct 3D workflow is used. The findings emphasize the importance of integrating intraoral scans early in the design stage to avoid errors in transverse dimensions. While limited by small sample size, this investigation provides foundational evidence for digital workflows and supports further research in larger populations.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years
* Good general health
* Satisfactory periodontal condition
* Proper oral hygiene
* Dissatisfaction with anterior maxillary esthetics
* Presence of complete maxillary anterior dentition without extensive restorations or severe discoloration

Exclusion Criteria:

* Active caries
* Untreated periodontal disease
* Missing teeth in the maxillary anterior region
* Severe malocclusion
* Poor oral hygiene

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Mesiodistal widths of anterior teeth - Comparison between digital designs and fabricated restorations. | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Incisogingival lengths of central and lateral incisors - Comparison between digital designs and fabricated restorations. | through study completion, an average of 1 year
Intercanine distance - Comparison between digital designs and fabricated restorations. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No